CLINICAL TRIAL: NCT04705714
Title: Antibacterial Activity of Boswellia Sacra Flueck. Oleoresin Extract Against Porphyromonas Gingivalis Periodontal Pathogen.
Brief Title: Antibacterial and Anti-biofilm Activity of Frankincense Extract Against Porphyromonas Gingivalis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, associate prof., Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2
Record Dates: First submitted 2021-01-03; First posted 2021-01-12 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Periodontal Diseases
Keywords: frankincense extract,; P. gingivalis ,; antibacterial activity;; susceptibility test of anaerobes; ; natural materials
MeSH Terms: conditions — Periodontal Diseases | interventions — Frankincense

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frankincense Extract (Experimental): the anti-bacterial and antibiofilm activity of frankincense extract against Porphyromonas gingivalis clinical isolates were studied
  Interventions: Drug: Frankincense Extract

INTERVENTIONS:
Drug: Frankincense Extract — The phytochemical composition of the volatile components of the extract was identified by GC-MS analysis, Crystal violet assay to test inhibition of biofilm formation by the tested isolates,Light microscope and scanning electron microscope were used to examine the biofilms and they confirmed the reduction of biofilm formation by frankincense extract
  Other Names: Boswellia sacra Flueck. Oleoresin Extract

SUMMARY:
Boswellia sacra Flueck. oleoresin extract (frankincense) was traditionally used in the treatment of different diseases as respiratory, rheumatoid arthritis, and bacterial infections. Therefore, the antibacterial and antibiofilm activity of frankincense extract against Porphyromonas gingivalis periodontal pathogen clinical isolates were studied

DETAILED DESCRIPTION:
The study was carried out on 30 systemically healthy patients of both sexes their ages ranged from 25 to 50 years old, diagnosed with moderate to severe chronic periodontitis (grade III stage b periodontitis), and selected from the clinic of Periodontology, Faculty of Dentistry, Tanta University

Gingival crevicular fluid samples (GCF) were collected from pockets having ≥ 5 mm depth and positive bleeding on probing (active disease) with a paper point. Samples were obtained from the periodontal pockets after removing the supragingival plaque from the teeth to be sampled. The subgingival plaque samples were then inoculated into 2 ml brain heart infusion (BHI) broth supplemented with 5 μg/mL hemin and 1 μg/mL menadione (vitamin K1). They were then diluted and cultured onto blood agar supplemented with 5% sheep blood, hemin (5 μg/mL) and vitamin K1 (0.5 μg/mL). These plates were incubated in duplicate for 7-10 days at 37 °C in an anaerobic atmosphere. The bacteria grown were finally selected based on their color, size, and shape. The black-pigmented colonies and Gram-negative rods (when examined microscopically) were examined by a fluorescence test using longwave UV light. The absence of fluorescence distinguishes between P. gingivalis and other anaerobic, black-pigmented, Gram-negative rods. The identification of P. gingivalis isolates was then confirmed using API 20A (BioMérieux, France).

4.8. Antibacterial screening It was performed using the agar diffusion method [40]. In brief, bacterial suspension was distributed onto blood agar plate surfaces supplemented with 5% sheep blood, 1% (v/v) hemin, and 1% (v/v) vitamin K1, then sterilized 6 mm blank filter paper discs were impregnated with 25 µl of frankincense oleoresin extract with different concentrations ranging from 0.5 to 1000 µg/ml. Discs loaded with 10% DMSO was used as negative controls and tetracycline disc (30 µg) was used as a positive control. All Petri dishes were anaerobically incubated at 37°C for 48 hrs. Inhibition zone diameters were measured and the concentrations of frankincense extract which showed clear zones (inhibition zone) around the discs were regarded to have an inhibitory effect on the tested bacteria.

4.9. Determination of MIC values The MIC values of frankincense extract against P. gingivalis isolates were estimated using the broth microdilution method. Briefly, cultures of P. gingivalis were grown overnight in BHI broth containing hemin (5 µg/mL) and vitamin K1 (1 µg/mL). Then, 100 µL of bacteria plus 100 µL of serial dilutions (two-fold) of the frankincense extract (starting from 2000 µg/mL) in BHI were mixed in the wells of the microtitration plate. Each microtitration plate had a negative control well-containing BHI without bacteria and a positive control well containing only bacteria without the extract. After anaerobic incubation at 37°C for 24 hrs., bacterial growth was inspected visually. The MIC values were recorded as the lowest concentrations that caused an inhibition of the bacterial growth. All the following experiments were performed before and after treatment of P. gingivalis isolates with sub-inhibitory concentrations (0.5 MIC) of the frankincense extract.

4.10. Bacterial growth curve P. gingivalis isolates were cultured in blood agar plates, supplemented with 5% sheep blood, hemin (5 μg/mL), and vitamin K1 (0.5 μg/mL), for 5-7 days under anaerobic conditions at 37°C [43]. Then, a single colony of each isolate was inoculated into BHI broth, containing hemin (5 µg/mL) and vitamin K1 (1 µg/mL), and grown anaerobically for 24 hrs. The optical density (OD) values at 600 nm were detected every 2 hrs. using UV-VIS spectrophotometer (Shimadzu, Japan), and the growth curves were constructed via plotting the log OD against the sampling time (hrs.).

4.11. Measurement of nucleic acid leakage The release of nucleic acids from the bacterial cells was measured as described previously. P. gingivalis isolates, at log phase, were centrifuged and the pellets were resuspended in phosphate-buffered saline (PBS), and incubated under anaerobic conditions. The release of cellular nucleic acids was measured at different times of 0, 1, 2, and 4 hrs. through measuring the absorbance at 260 nm using an 1800 UV-VIS spectrophotometer (Shimadzu, Japan).

4.12. Antibiofilm activity of frankincense extract

It was performed as previously described . Briefly, 100 µL of P. gingivalis suspensions were inoculated and cultured into a 96 well microtitration plate at anaerobic conditions at 37 °C. After incubation for 72 hrs., the non-adherent cells were removed via washing with PBS, and they were left to dry for 1 hr. The biofilms were stained using a solution of 0.1% crystal violet and the samples were washed with distilled water. For quantitative analysis of biofilm production, 125 µL of 30% acetic acid was added and the OD at 492 nm was measured using ELISA Auto Reader (Sunrise Tecan, Austria). The percentage of biofilm reduction was calculated using the formula:

% reduction of biofilm formation=(OD untreated-OD treated)/(OD untreated) x 100 Measurement of the extracellular polysaccharides The polysaccharides found in the extracellular polymeric substance (EPS) of the formed biofilm were estimated using the phenol-sulfuric acid method [43]. In brief, microtitration plates, after 3 days of biofilm formation by P. gingivalis isolates, were washed with PBS to remove the free-floating bacteria and air-dried. Then, 40 µL sterile water plus 40 µL 6% phenol solution, followed by 200 µL 97% sulfuric acid was added to each well. The plates were then left at room temperature for 30 min and the number of polysaccharides in the formed biofilm were determined by measuring the absorbance at an OD of 490 nm using ELISA Auto Reader (Sunrise Tecan, Austria). We used different glucose concentrations (0, 5, 10, 20, and 100 mg/L) as a standard to convert the OD values to polysaccharide concentrations.

4.14. Bacterial cell surface hydrophobicity

The bacterial hydrophobicity was assessed using the hydrocarbon-xylene test. Briefly, P. gingivalis isolates were cultured anaerobically and the pellets collected after centrifugation were resuspended in phosphate urea magnesium sulfate buffer (PUM buffer, pH 6.9). Then, volumes of 0.3, 0.9, 1.2, and 1.8 ml of n-hexane were added to 4.8 ml of the bacterial suspension. The mixtures were left for 2 hrs and the aqueous phase was cautiously separated. The absorbance of the tested isolates that remained in the aqueous phase was measured at 540 nm. HI was identified by the following equation:

HI=(A540 control-A540 test)/(A540 control) 4.15. Examination of biofilm morphology by light microscope and SEM It was carried out according to Qi et al. Briefly, two groups of glass cover slides were flooded with P. gingivalis isolates (with and without frankincense extract) and they were left for three days under anaerobic conditions to allow the isolates to form biofilms. The first group of the formed biofilms by P. gingivalis isolates was visualized by a bright-field microscope (Labomed, America) using 100× magnification after staining with crystal violet. The second group of the formed biofilms was rinsed using PBS and submerged in 2.5% glutaraldehyde solution for 24 hrs at 4°C. Then, they were sequentially dehydrated using a series of ethanol; concentrations ranging from 30% to 100%, let to dry, and sputter-coated with gold for examination with SEM (Hitachi, Japan).

4.16. qRT-PCR Relative gene expression of fimA, hagA, hagB, rgpA and kgp genes was examined using qRT-PCR. The used primers are listed in Table S1 and the 16S rRNA gene was the housekeeping gene or endogenous control. All the experiments were performed three times and the results values were expressed as mean ± standard deviation (SD). The amplification was carried out by Power SYBR® Green master mix (Thermo SCIENTIFIC, USA) using Rotor-Gene Q5 plex instrument (Qiagen, Germany). The relative gene expression was determined using the method of 2-ΔΔCt using the untreated isolates as control samples (its expression was set to 1). Changes in the gene expression with ≥ 2-fold (increased or decreased) were considered to be statistically significant

ELIGIBILITY:
Inclusion Criteria:

* patients with grade III stage b periodontitis , patients who have the willing to participate in the study and informed consents will be taken from them

Exclusion Criteria:

* patients who are under antibiotic therapy or any antimicrobial drugs
* smokers

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
isolation of the p. gingivalis | at day zero for in vitro study
  Isolated bacteria will be cultured on specific media and Antimicrobial activity of the extract will be examined by disc diffusion method

SECONDARY OUTCOMES:
GC-MS analysis | "up to 24 weeks"
  The phytochemical composition of the volatile components of the extract was identified by GC-MS analysis

OTHER OUTCOMES:
Crystal violet assay | baseline
  Crystal violet assay to test inhibition of biofilm formation by the tested isolate
Light microscope and scanning electron microscope | "up to 24 weeks"
  Light microscope and scanning electron microscope were used to examine the biofilms and they confirmed the reduction of Light microscope and scanning electron microscope were used to examine the biofilms and they confirmed the reduction of biofilm formation by frankincense extract biofilm formation by frankincense extract
qRT-PCR | "up to 24 weeks"
  Downregulation of the genes linked to biofilm formation (fimA, hagA, and hagB) was observed using qRT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: malak m shoukheba, PHD, Principal Investigator — faculty of dentistry tanta university
Locations (1):
- Malak Mohamed Shoukheba, Tanta, Egypt